CLINICAL TRIAL: NCT01578330
Title: A 12 -Month, Open-label, Multi-center Pilot Study to Explore the Health Outcomes of FTY720 in RRMS Patients Who Have Previously Been Treated With Other Disease Modifying Therapies (DMT)- Fine
Brief Title: A 12 -Month, Open-label, Multi-center Study to Explore the Health Outcomes of FTY720
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CFTY720DTR01
Record Dates: First submitted 2012-03-16; First posted 2012-04-16 (Estimated); Results first posted 2016-06-07 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-04

CONDITIONS: Multiple Sclerosis; Relapsing-Remitting
Keywords: Relapsing remitting multiple sclerosis; Fingolimod; FTY720
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting | interventions — Fingolimod Hydrochloride

ARMS (1):
- Fingolimod, FTY720 (Experimental): Patients received fingolimod 0.5 mg oral capsules daily with or without food.
  Interventions: Drug: Fingolimod

INTERVENTIONS:
Drug: Fingolimod — Fingolimod 0.5mg orally once a day without food.

SUMMARY:
The study will assess the patients' satisfaction of treatment after 12 months treatment with fingolimod It also will assess the tolerability profile of fingolimod in a small population.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with RRMS as described in 2005 Mc Donald criteria
2. Provided written informed consent prior to any intervention
3. Female or male patients aged 18-65 years
4. Unresponsive to treatment with a beta interferon or glatiramer acetate for a minimum of one year at and at adequate dose and with high disease activity

   (Unresponsive patients: patients with no changes in relapses, increased relapses, severer relapses with one-year treatment or those who had had at least one relapse during the past one year under previous treatments and one or multiple contrast enhancing lesions in cranial MRI or increased T2 lesions in successive MRIs)
5. EDSS score below 5.5 at baseline

Exclusion Criteria:

* Treatment-naive RRMS patients 2. History of a chronic disease of the immune system other than MS or known immunodeficiency 3. Past or current malignancy 4. Diabetic patients with mild or severe, non-proliferative or proliferative diabetic retinopathy and uncontrolled diabetic patients with HbA1c > 8% 5. Evidence of macular edema (patients with a history of macular edema will be allowed to enter the study provided that they do not have macular edema at screening.) 6. Evidence of uveitis 7. EDSS score > 5.5 at baseline 8. Active systemic bacterial, viral or fungal infections, or known to have AIDS, Hepatitis B, Hepatitis C infection or have positive HIV antibody, Hepatitis B surface antigen or Hepatitis C antibody tests 9. No history of varicella and negative varicella-zoster virus IhH antibody test at screening (such patients may be included after being administered VZV vaccine, at least 1 month following vaccination.) 10. Patients who received any live or live attenuated vaccine during the last one month (including varicella-zoster virus or measles) 11. Patients who received total lymphoid irradiation or bone marrow transplantation 12. Patient who received any of the treatment below:

  1. Corticosteroids or adrenocorticotropic hormone (ACTH) during the last 1 month
  2. Immunosuppressive medications such as azathioprine or methotrexate etc.
  3. Immunoglobulin treatment during the last 3 months
  4. Cladribine, cyclophosphamide, mitoxantrone, natalizumab at any time 13. Patients with any of the following cardiovascular conditions: Resting heart rate < 45 bpm/min Cardiac failure at time of screening (Class III according to NYHA classification) or any severe cardiac as determined by the physician Myocardial infarction during the last 6 months History of Mobitz Type II grade 2 AV block Past or current grade 3 AV block Confirmed history of sick sinus syndrome or sino-atrial heart block arrhythmia requiring current treatment with Class Ia drugs (ajmaline, disopyramid, procainamide, quinidine) hypertension uncontrolled with medication 14. Patients with any of the pulmonary conditions below severe respiratory disease or pulmonary fibrosis Uncontrolled asthma 15. Pregnant or nursing (lactating) women (pregnancy is defined as the state of a female after conception and until the termination of gestation and should be confirmed by a positive hCG laboratory test (> 5 mIU/ml).

     16. Patients with any of the hepatic conditions below: Alcohol abuse, chronic hepatic or biliary disease, severe hepatic impairment (Child- Pugh class C) Total bilirubin above the upper limit of normal provided that it is not associated with Gilbert's syndrome Conjugated bilirubin above the upper limit of normal Alkaline phosphate (AP) 1.5 times above the upper limit of normal AST(SGOT), ALT (SGPT) 2 times above the upper limit of normal, gamma-glutamyl-transferase (GGT) 3 times above the upper limit of normal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- Turkey (Türkiye) (10):
  - Novartis Investigative Site, Ankara, Turkey
  - Novartis Investigative Site, Bursa, Turkey
  - Novartis Investigative Site, Izmir, Turkey
  - Novartis Investigative Site, Altunizade
  - Novartis Investigative Site, Atakum / Samsun
  - Novartis Investigative Site, Fatih / Istanbul
  - Novartis Investigative Site, Kocaeli
  - Novartis Investigative Site, Mecidiyekoy/Istanbul
  - Novartis Investigative Site, Trabzon
  - Novartis Investigative Site, Uskudar / Istanbul

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fingolimod, FTY720
Started | 42
Per Protocol Population | 35
Completed | 35
Not Completed | 7
Not completed — Adverse Event | 2
Not completed — Protocol Violation | 5

BASELINE CHARACTERISTICS:
Arm/Group | Fingolimod, FTY720
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.7 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Mean Patient-Reported Treatment Satisfaction Questionnaire for Medication Scores (TSQM-9)
Description: The Treatment Satisfaction Questionnaire for Medication (TSQM-9) is a psychometric measure of a patient's satisfaction with medication. It consists of 3 subscales: effectiveness, convenience and global satisfaction. The scores were computed by adding items for each domain, i.e. 1 to 3 for effectiveness, 4 - 6 for convenience and 7 to 9 for global satisfaction. The lowest possible score (1 for each item and 3 for all 3 subscales) was subtracted from the composite score and divided by the greatest possible score range. The greatest range was (7-1) X 3 items = 18 for the effectiveness and convenience, and (5-1) x 3 items = 12 for global satisfaction. This provided a transformed score between 0 and 1 that was then multiplied by 100. A positive change from baseline indicates improvement.
Time Frame: Baseline and month 12
Population: Per Protocol Population: included all patients who had evaluable data for the primary variable from first to last visit
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Fingolimod, FTY720
Number analyzed (Participants) | 35
Scores on a scale
  Baseline (n=34) | 32.0 (9.9)
  Month 12 (n=32) | 44.7 (9.9)

2. Secondary Outcome: Mean Patient-reported Health-related Quality-of-life With Fingolimod (Short Form Health Survey: SF-36).
Description: The SF-36v2 is a validated health-related quality of life instrument used in numerous disease states, including MS. It is a self-administered survey that measures 8 domains of health including: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems and general mental health. Additionally, two summary scale scores can be calculated: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). If half or more questions within a domain were answered, then a score was calculated for that domain. Otherwise, the patient score for that domain was set to missing. If the patient was missing any 1 of the 8 scale scores, then the physical and mental component scores were set to missing. An algorithm was used to create a score from 0 to 100 for each domain score and component score. A positive change from baseline indicates improvement.
Time Frame: Month 1
Population: Per Protocol Population: included all patients who had evaluable data for the primary variable from first to last visit
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Fingolimod, FTY720
Number analyzed (Participants) | 35
score on scale
  Physical Function | 59.7 (30.9)
  Physical Role | 53.6 (43.8)
  Pain | 61.7 (23.7)
  General Health | 47.8 (20.5)
  Vitality | 28.9 (23.1)
  Social Function | 61.8 (26.4)
  Emotional Role | 48.4 (43.0)
  Mental Health | 31.5 (17.0)

3. Secondary Outcome: Mean Patient-reported Health-related Quality-of-life With Fingolimod (Short Form Health Survey: SF-36).
Description: as for outcome 2
Time Frame: Month 6
Population: Per Protocol Population: included all patients who had evaluable data for the primary variable from first to last visit
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Fingolimod, FTY720
Number analyzed (Participants) | 35
score on scale
  Physical Function (n=33) | 57.9 (31.1)
  Physical Role (n=34) | 47.8 (46.0)
  Pain (n=34) | 62.6 (24.8)
  General Health (n=33) | 48.5 (20.3)
  Vitality (n=34) | 35.2 (22.9)
  Social Function (n=34) | 60.6 (29.9)
  Emotional Role (n=34) | 54.8 (43.3)
  Mental Health (n=34) | 36.5 (20.3)

4. Secondary Outcome: Mean Patient-reported Health-related Quality-of-life With Fingolimod (Short Form Health Survey: SF-36).
Description: as for outcome 2
Time Frame: Month 12
Population: Per Protocol Population: included all patients who had evaluable data for the primary variable from first to last visit
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Fingolimod, FTY720
Number analyzed (Participants) | 35
score on scale
  Physical Function (n=31) | 59.5 (34.3)
  Physical Role (n=32) | 46.9 (44.7)
  Pain (n=32) | 65.9 (23.3)
  General Health (n=31) | 50.8 (21.9)
  Vitality (n=32) | 33.1 (20.0)
  Social Function (n=32) | 65.8 (29.1)
  Emotional Role (n=31) | 52.7 (46.2)
  Mental Health (n=32) | 36.3 (20.3)

ADVERSE EVENTS:
Arm/Group | Fingolimod, FTY720
Serious Adverse Events (participants affected / at risk) | 4/42
Other Adverse Events (participants affected / at risk) | 24/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod, FTY720 (N=42)
Multiple Sclerosis aggravated (Immune system disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Medication taken before pregnancy (Injury, poisoning and procedural complications) | 1
Middle ear infection surgery (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod, FTY720 (N=42)
Urinary infection (Renal and urinary disorders) | 9
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 8
Increase of hepatic enzymes (Hepatobiliary disorders) | 5
Lymphopenia (Blood and lymphatic system disorders) | 7
Multiple Sclerosis Aggravated (Immune system disorders) | 4
Headache (Nervous system disorders) | 4
Hyperlipidemia (Metabolism and nutrition disorders) | 4
Tooth abscess (Infections and infestations) | 3
Nausea (Gastrointestinal disorders) | 3
Incontinence (Renal and urinary disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety